CLINICAL TRIAL: NCT03206437
Title: Effect of Mindfulness Meditation on Physiological Response to Unpredictable Stimuli
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Georgetown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2017-0698
Record Dates: First submitted 2017-06-28; First posted 2017-07-02 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-12

CONDITIONS: Anxiety Disorders; Generalized Anxiety Disorder; Social Anxiety Disorder; Panic Disorder; Post Traumatic Stress Disorder; Agoraphobia; Simple Phobia
Keywords: mindfulness; meditation
MeSH Terms: conditions — Anxiety Disorders; Generalized Anxiety Disorder; Phobia, Social; Panic Disorder; Stress Disorders, Post-Traumatic; Agoraphobia; Phobia, Specific | interventions — Mindfulness-Based Stress Reduction; Waiting Lists

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: Since this study is focusing on a mind-body skill as a treatment it will be impossible to mask the participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness-Based Stress Reduction (Experimental): This group will take the 8 week MBSR course within 4 weeks of their first testing visit. When the course is finished they will come in for their second testing visit. The course meets once a week in person for 2.5 hours and participants are expected to do practices at home.
  Interventions: Behavioral: Mindfulness-Based Stress Reduction
- Waitlist (Other): The wait-list group will not participate in the MBSR course within 4 weeks of their first testing visit. They will wait 8-16 weeks and come on for a second testing visit. After their data is collected they will be offered an MBSR course to take.
  Interventions: Behavioral: Waitlist

INTERVENTIONS:
Behavioral: Mindfulness-Based Stress Reduction — The MBSR course teaches mindfulness meditation skills. This 8-week course meets in person once a week for 2.5 hours. Participants are expected to complete practice assignments at home.
  Arms: Mindfulness-Based Stress Reduction
Behavioral: Waitlist — This group will wait 8-16 weeks after their first testing visit and after their second study visit is completed they will be able to participate in an 8-week MBSR course.
  Arms: Waitlist

SUMMARY:
This study will evaluate the effects of Mindfulness-Based Stress Reduction (MBSR) on physiological reactivity. This study will focus on individuals with anxiety who will participate in an 8-week MBSR class. The investigators will test participants' reactivity to both predictable and unpredictable stimuli before and after the class to understand the physiological changes that may occur after to the intervention. Secondary measures include psychometric instruments and a delay discounting task.

DETAILED DESCRIPTION:
Mindfulness-Based Stress Reduction (MBSR) is a manualized, systematic training in mindfulness meditation that has been found to have beneficial health effects, such as decreased stress and anxiety. The current protocol aims to examine the effects of MBSR on several physiological and behavioral measures in people with anxiety disorders, which may help us understand the effects of the intervention on anxiety. The investigators will use the NPU task as developed by the NIH, which measures an individual's response to threatening stimuli (mild shock) paired with non-threatening stimuli (geometric shapes). Individuals with anxiety disorders will be recruited to participate in this study, and will be randomized to a control (waitlist) or MBSR intervention group. Other secondary measures will examine the effects of mindfulness meditation on decision-making, and stress and anxiety symptoms.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women from 18-65 years of age.
2. Have an anxiety disorder, including: social anxiety disorder (SAD), generalized anxiety disorder (GAD), panic disorder, posttraumatic stress disorder (PTSD), agoraphobia, or simple phobia.
3. Must understand study procedure and willing to participate in 2 testing visits, and MBSR course as assigned.
4. Participants must be able to give informed consent to the study procedures.

Exclusion Criteria:

1. Subjects experiencing a current depressive episode or other axis I psychiatric disorders such as psychotic disorders, obsessive compulsive disorder, current eating disorders, bipolar disorder, and current substance use disorders.
2. Lack of measurable eye blink/eye twitch response (3 times the baseline eye blink muscle activity as measured by electromyography) for at least 5 of 9 startles used during the habituation visit.
3. A serious medical condition that may result in surgery or hospitalization.
4. Subjects who will be non-compliant with the study procedures. This may include planned travel out of town.
5. Women who are pregnant.
6. Current evidence of median nerve entrapment or carpal tunnel syndrome.
7. Subject who has resting blood pressure outside of a systolic blood pressure range of 90-140 mmHg, or a diastolic blood pressure outside a range of 50-90 mmHg on two consecutive measurements, taken up to 10 minutes apart.
8. Subjects taking benzodiazepines, barbiturates, antidepressants, antipsychotics, or sedative medications
9. Subjects currently receiving concomitant psychotherapy directed at treating anxiety symptoms (i.e. CBT).
10. Individuals with implanted electronic devices, such as a cardiac pacemaker.
11. Individuals who have completed a full course of MBSR, an equivalent meditation training, or have a daily meditation practice.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2017-06-20 (Actual); Primary Completion 2022-11-25 (Actual); Study Completion 2022-11-25 (Actual)

PRIMARY OUTCOMES:
Fear and anxiety potentiated startle | 16 weeks
  This variable will be measured by using the Neutral, Predictable, and Unpredictable (NPU) Threat Test

SECONDARY OUTCOMES:
Center for Epidemiologic Studies Depression Scale (CES-D), | 16 weeks
  measures depression symptoms
The State-Trait Anxiety Inventory (STAI) | 16 weeks
  This is a measure of state and trait anxiety
Delay Discounting | 16 weeks
  This is a computer task that measures a decline in reward value over a given time

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Hoge, Principal Investigator — Georgetown University
Locations (1):
- Georgetown University Medical Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schmitz A, Grillon C. Assessing fear and anxiety in humans using the threat of predictable and unpredictable aversive events (the NPU-threat test). Nat Protoc. 2012 Feb 23;7(3):527-32. doi: 10.1038/nprot.2012.001. PMID 22362158